CLINICAL TRIAL: NCT00925951
Title: The Effectiveness of Wet Cupping on Persistent Non-specific Low Back Pain: A Randomized, Waiting-list Controlled, Open-label, Parallel-group Pilot Study
Brief Title: The Effectiveness of Wet Cupping on Persistent Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Kim Ki-ok, Korea Institute of Oriental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI0905
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-06

CONDITIONS: Low Back Pain
Keywords: Persistent Non-specific Low Back Pain; wet cupping; cupping; Numerical Rating Scale
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wet Cupping (Experimental)
  Interventions: Device: Wet Cupping; Drug: Acetaminophen
- Waiting Control (No Intervention): They can't use any other specific treatment except exercises and behavior modification (we'll offer a brochure which includes exercise method and directions about behavior modifications).
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Device: Wet Cupping — Wet cupping (Seongho trade & company, Korea) will be practiced at two selected points (among the 6 acupoints, left or right BL23, BL24, BL25)
  Other Names: Disposable wet cupping cup, Seongho trade & company, Korea
  Arms: Wet Cupping
Drug: Acetaminophen — Acetaminophen 500 mg tablets will be offered to both of the wet cupping group and waiting group for relieving severe pain.

SUMMARY:
The hypothesis of this study is that the improvement of Numeric Rating Scale (NRS) for Pain at the end of the study will be greater in the Wet Cupping Treatment group than in the Waiting Control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had non-specific low back pains at least 12 weeks now.

Exclusion Criteria:

* Patients who have low back pain due to specific and known etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome, cauda equinal syndrome).
* Patients who are inappropriate to the wet cupping treatment.

  * AIDS, Active Hepatitis, Tuberculosis, Syphilis
  * Patients who regularly take anticoagulants, antiplatelet drugs
  * Anemia, thrombocytopenia
  * Hemorrhagic disease like hemophilia
  * Diabetes
  * Severe cardiovascular disease
  * Kidney diseases (renal failure, chronic renal disease)
* Patients who have experiences of wet cupping treatment during last 3 months.
* Patients who have had treatment for low back pain during last 2 weeks.
* Patients who are in pregnancy or have plan to conception.
* Patients who have vertebra surgery or have plan of surgery.
* Patients who are inappropriate to join this trial judged by the radiologists or specialists.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) for pain | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation

SECONDARY OUTCOMES:
Present Pain Intensity Scale of the McGill Pain Questionaire (PPI) | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation
Oswestry Disability Questionnaire (ODQ) | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation
Medication Quantification Scale (MQS) | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation
General Assessment of Doctors and Subjects | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation
Safety measurement | study group: at base line, post-treatment, 4 weeks later after allocation; control group: at base line, 4 weeks later after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Sun-mi Choi, Doctor, Study Chair — Korea Institute of Oriental Medicine (KIOM); Jong-In Kim, Doctor, Study Director — Korea Institue of Oriental Medicine (KIOM); Tae-hun Kim, Doctor, Principal Investigator — Korea Institue of Oriental Medicine (KIOM)
Locations (1):
- Korea Institue of Oriental Medicine (KIOM), Doonsan Oriental Hospital of Daejeon University, Daejeon, Chungchong, South Korea

REFERENCES:
- [Derived] Kim JI, Kim TH, Lee MS, Kang JW, Kim KH, Choi JY, Kang KW, Kim AR, Shin MS, Jung SY, Choi SM. Evaluation of wet-cupping therapy for persistent non-specific low back pain: a randomised, waiting-list controlled, open-label, parallel-group pilot trial. Trials. 2011 Jun 10;12:146. doi: 10.1186/1745-6215-12-146. PMID 21663617